CLINICAL TRIAL: NCT02407951
Title: Tel Aviv Sourasky Medical Center
Brief Title: Group Intervention for Children With Chronic Tics Syndrome or Tourette Syndrome: CBIT vs Psycho-Educational Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0437-17-TLV
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Tourette Syndrome; Motor or Vocal Tic Disorder, Chronic
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBIT group (Experimental)
  Interventions: Behavioral: CBIT group
- Psycho-Educational group (Placebo Comparator)
  Interventions: Behavioral: Psycho-Educational group

INTERVENTIONS:
Behavioral: CBIT group — Child group: 8 weekly group sessions lasting 90 mins, additional three monthly booster sessions.
  During sessions, children create a tic hierarchy from most to least distressing, with more distressing tics addressed earlier in the treatment. Awareness training and competing response training is implemented and practiced. Competing response training is added, involving engagement in a voluntary behavior physically incompatible with the tic, contingent on the premonitory urge or other signs of impeding tic occurrence. Relaxation training addresses situations that sustained or worsened tics, training focuses on developing individual behavioral strategies to reduce the influence of these factor.
  Parallel parent-group sessions simultaneously run during first 4 sessions of child-group. parents-group includes psycho-education and use of reward strategies.
  Meetings executed by two trained clinicians.
  Arms: CBIT group
Behavioral: Psycho-Educational group — Child group: 8 weekly group sessions lasting 90 mins each, as well as additional three monthly booster sessions afterwards.
  During the educational group sessions, each session will focus on educating the participants in regard to a specific subject: Tourette syndrome, Self-esteem, Anger, OCD (obssesive compulsive disorder), School and bullying, Anxiety, Attention, and a final session Quiz.
  Parent group: Parent-group sessions will simultaneously run during the first 4 sessions of the child-group. The parents-group will include psycho-education and the use of reward strategies.
  All group meetings will be executed and managed by two trained clinicians.
  Arms: Psycho-Educational group

SUMMARY:
Tourette Syndrome (TS) is a disorder characterized by motor and vocal tics. The most studied and promising intervention is Habit Reversal Training (HRT) and its variations: Behavioral Comprehensive Intervention for Tics (CBIT). Group intervention for children with TS has not been evaluated. The aim of this study is to assess the efficacy of CBIT group intervention compared with Psycho-Educational-Supportive group in terms of tic severity.

DETAILED DESCRIPTION:
Tourette Syndrome (TS) is a neuro-developmental disorder characterized by motor and vocal tics, frequently associated with behavioral and functional problems, impacting significantly on children's quality of life . Current evidence supports the contribution of individual behavioral treatment for TS both for reducing tics and improving children's quality of life. The most studied and promising intervention is Habit Reversal Training (HRT) and its variations: Behavioral Comprehensive Intervention for Tics (CBIT). One of the developments of behavioral treatments is group interventions, supported in various types of psychological difficulties, adding benefit of providing peer support. However, group intervention for children with TS has not been empirically evaluated.

The aim of this study is to assess the efficacy of CBIT group intervention. We hypothesize that CBIT group intervention will be more effective than Psycho-Educational-Supportive (PES) group in terms of tic severity, and that both groups will be effective in quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Tourettes syndrome or chronic tic disorder
* age 9-15 years
* native Hebrew speakers

Exclusion Criteria:

* intellectual disability (FSIQ < 80)
* current diagnosis of substance abuse/dependence
* life time diagnosis of pervasive developmental disorder, mania or psychosis.
* previous treatment with 4 or more individual sessions of CBIT

Children receiving medications for tics: eligible if the dose is stable for 6 weeks prior to study with no planned changes during study participation.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale | 3 months
  semi-structured clinical interview carried out with parent and child. Questions relate to tic severity over the previous week. Separate ratings are recorded for motor and phonic tics in terms of their number, frequency, intensity, complexity, and interference on a 6-point Likert scale. Three composite scores are generated which are total motor tic severity (rated from 0 to 25), total phonic tic severity (rated from 0 to 25) and total tic severity overall (rated from 0 to 50).

REFERENCES:
- [Background] Woods DW, Piacentini JC, Scahill L, Peterson AL, Wilhelm S, Chang S, Deckersbach T, McGuire J, Specht M, Conelea CA, Rozenman M, Dzuria J, Liu H, Levi-Pearl S, Walkup JT. Behavior therapy for tics in children: acute and long-term effects on psychiatric and psychosocial functioning. J Child Neurol. 2011 Jul;26(7):858-65. doi: 10.1177/0883073810397046. Epub 2011 May 9. PMID 21555779
- [Derived] Zimmerman-Brenner S, Pilowsky-Peleg T, Rachamim L, Ben-Zvi A, Gur N, Murphy T, Fattal-Valevski A, Rotstein M. Group behavioral interventions for tics and comorbid symptoms in children with chronic tic disorders. Eur Child Adolesc Psychiatry. 2022 Apr;31(4):637-648. doi: 10.1007/s00787-020-01702-5. Epub 2021 Jan 7. PMID 33415472